CLINICAL TRIAL: NCT03010176
Title: Phase 1 Open-label, Multicenter Study of MK-1454 Administered by Intratumoral Injection as Monotherapy and in Combination With Pembrolizumab for Patients With Advanced/Metastatic Solid Tumors or Lymphomas
Brief Title: Study of Ulevostinag (MK-1454) Alone or in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic Solid Tumors or Lymphomas (MK-1454-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1454-001; MK-1454-001 (Other: Merck); 2016-003160-40 (EudraCT Number)
Record Dates: First submitted 2017-01-03; First posted 2017-01-04 (Estimated); Results first posted 2024-02-26 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors; Lymphoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Intratumoral (IT)
MeSH Terms: conditions — Lymphoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) (Experimental): Participants with cutaneous (cut) or subcutaneous (subcut) lesions will receive escalating doses of ulevostinag monotherapy via IT injection on Days 1, 8, and 15 of each 21-day cycle for Cycles 1, 2, and 3 and then on Day 1 of each 21-day cycle for Cycles 4 and beyond for up to 35 cycles (up to approximately 2 years).
  Interventions: Drug: Ulevostinag
- Part 1 Arm 2: Ulevostinag +Pembro (Cut/Subcut Lesions) (Experimental): Participants with cut or subcut lesions will receive escalating doses of ulevostinag via IT injection on Days 1, 8, and 15 of each 21-day cycle for Cycles 1, 2, and 3 and then on Day 1 of each 21-day cycle for Cycles 4 and beyond PLUS pembrolizumab (pembro) via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Drug: Ulevostinag; Biological: Pembrolizumab
- Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) (Experimental): Participants with visceral lesions will receive escalating dose frequencies of ulevostinag via IT injection at escalating dose frequencies (Day 1 of each 21-day cycle for up to 35 cycles, then Days 1 and 8 of each 21-day cycle for two cycles, then Day 1 of each 21 day cycle up to 35 cycles, then Days 1, 8, and 15 of each 21-day cycle for two cycles followed by Day 1 of each 21-day cycle up to 35 cycles, PLUS pembrolizumab IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (approximately 2 years).
  Interventions: Drug: Ulevostinag; Biological: Pembrolizumab
- Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory (Experimental): Participants with HNSCC who are anti-programmed cell death-1 or anti-programmed cell death-ligand 1 refractory will receive ulevostinag at the preliminary Recommended Phase 2 Dose (RP2D) determined by dose escalation in Part 1 Arm 1 and 2 via IT injection on Days 1, 8, and 15 of Cycles 1 and 2 and on Day 1 of each 21-day cycle from Cycle 3 onward (up to a total of 35 cycles) PLUS pembrolizumab via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Drug: Ulevostinag; Biological: Pembrolizumab
- Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC (Experimental): Participants with TNBC who are anti-PD-1/PD-L1 treatment-naïve or who have refractory unresectable locally advanced or metastatic TNBC will receive ulevostinag at the preliminary RP2D determined by dose escalation in Part 1 via IT injection on Days 1, 8, and 15 of Cycles 1 and 2 and on Day 1 of each 21-day cycle from Cycle 3 onward (up to a total of 35 cycles) PLUS pembrolizumab via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Drug: Ulevostinag; Biological: Pembrolizumab
- Part 2 Cohort C: Anti-PD-1/PD-L1 TrT-Naïve Solid Tumors-Liver (Experimental): Participants with solid tumors with liver metastases/lesions who are anti-PD-1/PD-L1 treatment-naïve will receive ulevostinag at the preliminary RP2D based on Part 1: ulevostinag + pembro (visceral lesions) treatment arm via IT injection in a to-be-determined dose and frequency, based on data from Arm 3, PLUS pembrolizumab via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Drug: Ulevostinag; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Ulevostinag — IT injection
  Other Names: MK-1454
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; Keytruda®
  Arms: Part 1 Arm 2: Ulevostinag +Pembro (Cut/Subcut Lesions); Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions); Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory; Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC; Part 2 Cohort C: Anti-PD-1/PD-L1 TrT-Naïve Solid Tumors-Liver

SUMMARY:
The purpose of this study is to identify a maximum tolerated dose (MTD) or maximum administered dose (MAD) of ulevostinag alone and of ulevostinag in combination with pembrolizumab in participants with advanced/metastatic solid tumors or lymphomas in Part 1, and to evaluate the safety and efficacy of ulevostinag via intratumoral (IT) injection in combination with pembrolizumab in selected solid tumors in Part 2.

Ulevostinag will be administered IT; pembrolizumab (pembro) will be administered via intravenous (IV) infusion. In Part 1, participants will be allocated to one of three treatment arms: ulevostinag monotherapy (cutaneous/subcutaneous [cut/subcut] lesions), ulevostinag +pembro (cut/subcut lesions), or ulevostinag +pembro (visceral lesions).

In Part 2, participants with head and neck squamous cell carcinoma (HNSCC) who are anti-programmed cell death-protein 1 or anti-programmed cell death-ligand 1 (anti-PD-1/PD-L1) refractory or with anti-PD-1/PD-L1 treatment (TrT)-naïve triple-negative breast cancer (TNBC) or with anti-PD-1/PD-L1 TrT-naïve solid tumors with liver metastases/lesions will receive ulevostinag via IT injection at the preliminary Recommended Phase 2 Dose (RP2D) determined in Part 1 PLUS pembrolizumab via IV infusion for up 35 cycles (up approximately 2 years).

DETAILED DESCRIPTION:
Participants will receive either ulevostinag monotherapy or ulevostinag in combination with pembrolizumab for up to 35 cycles (approximately 2 years). Participants will undergo at least a 24-hour inpatient observation period following the first dose administration of ulevostinag on Cycle 1 Day 1 in Part 1. For Part 2, the length of the observation period following administration of the first dose of ulevostinag on Cycle 1 Day 1 is at least 8 hours.

ELIGIBILITY:
Inclusion Criteria:

All Arms and Cohorts (Parts 1 and 2):

* Has ≥1 injectable lesion which is measurable and amenable to injection and biopsy.
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Demonstrates adequate organ function within 7 days prior to treatment initiation.
* Female participants of childbearing potential must be using a contraceptive method that is highly effective or be abstinent from heterosexual intercourse (on a long-term and persistent basis) during the intervention period and for at least 130 days after the last dose of study intervention and agrees not to donate eggs to others or freeze/store for personal use for the purpose of reproduction during this period. Male participants must agree to refrain from donating sperm PLUS either be abstinent from heterosexual intercourse (on a long-term and persistent basis) OR agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse contraception, unless confirmed to be azoospermic (vasectomized) during the intervention period and for at least 130 days after the last dose of study intervention.
* Human Immunodeficiency (HIV)-infected participants must meet these additional criteria: a) Has laboratory-test-documented HIV-1 infection; b) Has well-controlled HIV on anti-retroviral therapy (ART), defined as: 1) must have a cluster of differentiation (CD4+) T-cell count >350 cells/mm^3 at time of screening; 2) must have achieved and maintained virologic suppression defined as confirmed HIV ribonucleic acid (RNA) level below 50 or the lower limit of quantification (LLOQ) using the locally available assay at the time of screening and for ≥12 weeks prior to screening; and, 3) must have been on a stable regimen, without changes in drugs or dose modification, for ≥4 weeks prior to study entry (Day 1).

All Part 1 Arms:

-Has ≥1 distant, discrete non-injected lesion which is amenable to biopsy. This lesion must be measurable as defined by the response criteria used to assess the participant (RECIST 1.1 for solid tumors or revised International Working Group [IWG] criteria for lymphomas).

Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) and Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions):

* Has a histologically- or cytologically-confirmed advanced/metastatic solid tumor or lymphoma by pathology report and who has received, or been intolerant to, all treatment known to confer clinical benefit. Solid tumors and lymphomas of any type are eligible for enrollment.
* Has stage III or stage IV disease that is not surgically resectable. Stage IIB (T3N0M0B0-1) cutaneous T cell lymphoma (CTCL) participants are eligible.

Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions):

* Has stage III or stage IV disease that is not surgically resectable.
* Has metastatic liver involvement that does not exceed one third of the total liver volume in participants to be treated by liver IT injection. Hepatocellular carcinoma participants are excluded from eligibility of IT liver injection.

All Part 2 Expansion Cohorts:

Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory:

* Has HNSCC of the oral cavity, oropharynx, hypopharynx, or larynx; anti-PD-1/PD-L1 refractory metastatic or recurrent. Participants may not have a primary tumor site of the nasopharynx (any histology).
* Has histologically confirmed Stage III, IVa, or IVb disease per TNM (Tumor, Nodes, Metastasis) staging, American Joint Committee on Cancer (AJCC, 8th edition), with recurrent or persistent disease after definitive chemoradiation, deemed unresectable and considered refractory to both platinum-based combination chemotherapy and anti-programmed cell death-ligand 1 (anti-PD-1/PD-L1) antibody therapy.

OR

* Has histologically confirmed Stage IVc disease per TNM staging, AJCC 8th edition, considered refractory to platinum-based combination chemotherapy and anti-PD-1/PD-L1 antibody therapy.

Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC:

* Has confirmed unresectable locally advanced or metastatic TNBC as locally determined according to the American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) guidelines on a newly obtained core or excisional biopsy from a metastatic, not previously irradiated, tumor lesion.
* Has received at least one prior systemic treatment for metastatic breast cancer and has intolerance to, or documented disease progression on or after their most recent therapy.
* Has been previously treated with an anthracycline and/or taxane in the (neo)adjuvant or metastatic setting unless there was a medical contraindication to this treatment regimen.
* Have lactate dehydrogenase (LDH) <2.5 × upper limit of normal (ULN)

Part 2 Cohort C: Anti-PD-1/PD-L1 TrT-Naïve Solid Tumors-Liver:

* Has histologically or cytologically confirmed Stage IV solid tumor that is not surgically resectable.
* Complete resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or baseline (except alopecia). If participant received major surgery or radiation therapy of >30 Gray (Gy), they must have recovered from the toxicity and/or complications from the intervention.

Exclusion Criteria:

All Arms and Cohorts (Parts 1 and 2):

* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks prior to the first dose of study drug, or has not recovered to Baseline or Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 from the adverse events due to cancer therapeutics administered >4 weeks earlier.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and has received study therapy or has used an investigational device within 28 days of administration of ulevostinag. Note: Prior exposure to immunotherapeutics is allowed, including PD-1 and PD-L1 inhibitors
* Is expected to require any other form of antineoplastic therapy while on study.
* Is on chronic systemic steroid therapy in excess of replacement doses (prednisone ≤ 10 mg/day is acceptable), or on any other form of immunosuppressive medication.
* Has a history of a second malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for 2 years.
* Has clinically active central nervous system metastases and/or carcinomatous meningitis.
* Has had a severe hypersensitivity reaction to treatment with a monoclonal antibody.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has a history of vasculitis.
* Has an active infection requiring therapy.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years.
* Has Hepatitis B or C infection(s).
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Has not fully recovered from any effects of major surgery, and is free of significant detectable infection.
* Has received a live vaccine within 30 days prior to first dose of study drug.
* Has a history of re-irradiation for squamous cell carcinoma of the head & neck (HNSCC) at the projected injection site.
* Has a tumor(s) in direct contact or encases a major blood vessel, and has ulceration and/or fungation onto the skin surface at the projected injection site.
* HIV-infected participants with history of Kaposi's sarcoma and/or multicentric Castleman's disease
* HIV-infected participants who have had an HIV-related opportunistic infection within 6 months
* Has been treated with a Stimulator of Interferon Genes (STING) agonist (e.g. ulevostinag, ADU-S100).

All Part 2 Expansion Cohorts:

* Has experienced weight loss >10% over 2 months prior to first dose of study treatment.
* Has clinically relevant ascites at baseline (defined as requiring paracentesis) or with moderate radiographic ascites. A minimal amount of radiographic ascites is allowed.
* Has a history of interstitial lung disease.
* For Part 2 Cohort C: Anti-PD-1/PD-L1 TrT-Naïve Solid Tumors-Liver, participants with MSI-H CRC are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (19):
- United States (10):
  - University of Alabama ( Site 0009), Birmingham, Alabama
  - University of California San Francisco ( Site 0007), San Francisco, California
  - UCSF ( Site 0015), San Francisco, California
  - UCLA Medical Center ( Site 0005), Santa Monica, California
  - Henry Ford Health System ( Site 0014), Detroit, Michigan
  - Mount Sinai Hospital ( Site 0002), New York, New York
  - Columbia University ( Site 0003), New York, New York
  - UPMC Hillman Cancer Center ( Site 0013), Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research Center ( Site 0001), Dallas, Texas
  - Huntsman Cancer Institute ( Site 0004), Salt Lake City, Utah
- France (3):
  - Institut Claudius Regaud ( Site 0051), Toulouse, Haute-Garonne
  - Institut Gustave Roussy ( Site 0049), Villejuif, Val-de-Marne
  - Institut Curie ( Site 0050), Paris
- Israel (2):
  - Rambam Medical Center ( Site 0041), Haifa
  - Sheba Medical Center ( Site 0040), Ramat Gan
- South Korea (2):
  - Severance Hospital ( Site 0103), Seoul
  - Asan Medical Center ( Site 0104), Seoul
- United Kingdom (2):
  - The Royal Marsden Foundation Trust ( Site 0031), London, London, City of
  - The Royal Marsden NHS Foundation Trust. ( Site 0032), Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Harrington KJ, Champiat S, Brody JD, Cho BC, Romano E, Golan T, Hyngstrom JR, Strauss J, Oh DY, Popovtzer A, Gomez-Roca C, Perets R, Kim SB, Wong DJ, Powell SF, Khilnani A, Jemielita T, Zhao Q, Zhao R, Ingham M. Phase I and II Clinical Studies of the STING Agonist Ulevostinag with and without Pembrolizumab in Participants with Advanced or Metastatic Solid Tumors or Lymphomas. Clin Cancer Res. 2025 Aug 14;31(16):3400-3411. doi: 10.1158/1078-0432.CCR-24-3630. PMID 40499147
- [Derived] Gogoi H, Mansouri S, Jin L. The Age of Cyclic Dinucleotide Vaccine Adjuvants. Vaccines (Basel). 2020 Aug 13;8(3):453. doi: 10.3390/vaccines8030453. PMID 32823563

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Evaluation of Part 2 Cohort C (anti-PD-1/PD-L1 treatment-naïve solid tumors with liver metastases/lesions) was not pursued. No participants were enrolled in Part 2 Cohort C.
Groups:
- Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions): Participants with cutaneous (cut) or subcutaneous (subcut) lesions received escalating doses of ulevostinag monotherapy via intratumoral (IT) injection on Days 1, 8, and 15 of each 21-day cycle for Cycles 1, 2, and 3 and then on Day 1 of each 21-day cycle for Cycles 4 and beyond for up to 35 cycles (up to approximately 2 years).
- Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions): Participants with cut or subcut lesions received escalating doses of ulevostinag via IT injection on Days 1, 8, and 15 of each 21-day cycle for Cycles 1, 2, and 3 and then on Day 1 of each 21-day cycle for Cycles 4 and beyond PLUS pembrolizumab (pembro) via intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years).
- Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions): Participants with visceral lesions received escalating doses of ulevostinag via IT injection at escalating dose frequencies (Day 1 of each 21-day cycle for up to 35 cycles, then Days 1 and 8 of each 21-day cycle for two cycles, then Day 1 of each 21 day cycle up to 35 cycles, then Days 1, 8, and 15 of each 21-day cycle for two cycles followed by Day 1 of each 21-day cycle up to 35 cycles), PLUS pembrolizumab via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (approximately 2 years).
- Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory: Participants with head and neck squamous cell carcinoma (HNSCC) who were anti-programmed cell death-1 (anti-PD-1) or anti-programmed cell death-ligand 1 (anti-PD-L1) refractory received ulevostinag via IT injection on Days 1, 8, and 15 of Cycles 1 and 2 and on Day 1 of each 21-day cycle from Cycle 3 onward (up to a total of 35 cycles) PLUS pembrolizumab IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years).
- Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC: Participants with triple-negative breast cancer (TNBC) who were anti-PD-1/PD-L1 treatment (TrT)-naïve or who had refractory unresectable locally advanced or metastatic TNBC received ulevostinag via IT injection on Days 1, 8, and 15 of Cycles 1 and 2 and on Day 1 of each 21-day cycle from Cycle 3 onward (up to a total of 35 cycles) PLUS pembrolizumab via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years).
- Part 2 Cohort C: Anti-PD-1/PD-L1 TrT-Naïve Solid Tumors-Liver: Participants with solid tumors with liver metastases/lesions who were anti-PD-1/PD-L1 treatment-naïve were to receive ulevostinag at the preliminary RP2D based on Part 1: ulevostinag+pembro (visceral lesions) treatment arm via IT injection in a to-be-determined dose and frequency, based on data from Arm 3, PLUS pembrolizumab mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years).
Period: Overall Study
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC | Part 2 Cohort C: Anti-PD-1/PD-L1 TrT-Naïve Solid Tumors-Liver
Started | 32 | 52 | 26 | 21 | 25 | 0
Treated | 32 | 52 | 26 | 21 | 25 | 0
Switched From Part 1 Arm 1 to Part 1 Arm 2 (Switched over from Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) to Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions)) | 14 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 32 | 52 | 26 | 21 | 25 | 0
Not completed — Death | 21 | 35 | 19 | 19 | 14 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 4 | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 0 | 4 | 4 | 1 | 6 | 0
Not completed — Withdrawal by Subject | 11 | 9 | 3 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Evaluation of Part 2 Cohort C (anti-PD-1/PD-L1 treatment-naïve solid tumors with liver metastases/lesions) was not pursued. No participants were enrolled in Part 2 Cohort C.
Groups:
- Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions): Participants with cutaneous (cut) or subcutaneous (subcut) lesions received escalating doses of ulevostinag monotherapy via IT injection on Days 1, 8, and 15 of each 21-day cycle for Cycles 1, 2, and 3 and then on Day 1 of each 21-day cycle for Cycles 4 and beyond for up to 35 cycles (up to approximately 2 years).
- Total: Total of all reporting groups
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC | Part 2 Cohort C: Anti-PD-1/PD-L1 TrT-Naïve Solid Tumors-Liver | Total
Number analyzed (Participants) | 32 | 52 | 26 | 21 | 25 | 0 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (14.1) | 60.1 (14.0) | 59.1 (10.1) | 60.2 (8.5) | 49.3 (10.9) |  | 57.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 31 | 8 | 4 | 25 | 0 | 88
  Male | 12 | 21 | 18 | 17 | 0 | 0 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 30 | 44 | 25 | 20 | 12 | 0 | 131
  Unknown or Not Reported | 1 | 6 | 1 | 1 | 12 | 0 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 6 | 6 | 3 | 0 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 2 | 0 | 5
  White | 26 | 50 | 20 | 12 | 7 | 0 | 115
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 13 | 0 | 16

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Who Experienced a Dose-limiting Toxicity (DLT) Per Common Terminology Criteria for Adverse Events, Version 4.0 (CTCAE 4.0)
Description: DLTs were assessed during the first cycle (21 days) & are defined as: Grade (Gr) 4 nonhematologic toxicity; Gr 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia, Gr 4 thrombocytopenia, Gr 3 thrombocytopenia (if associated with clinically significant bleeding); nonhematologic adverse event (AE) ≥ Gr 3 (with exceptions); Gr 3 or 4 nonhematologic lab abnormality (if medical intervention is required, leads to hospitalization, or persists for >1 week); Gr 3 or 4 febrile neutropenia; drug-related toxicity that causes treatment discontinuation or dose delay >7 days between consecutive doses during Cycle 1; drug-related toxicity that causes a >2 week delay in Cycle 2 initiation; elevated aspartate aminotransferase or alanine aminotransferase lab value that is ≥3× upper limit of normal (ULN) & an elevated total bilirubin value ≥2× ULN & an alkaline phosphatase value <2× ULN, in which no alternative reasons can be found; ≥Gr 2 immune-mediated uveitis; or Gr 5 toxicity.
Time Frame: Cycle 1 (21-day cycle)
Population: All participants who received at least 1 dose of study treatment and were either observed for safety for 21 days after the first dose of treatment or experienced a DLT prior to 21 days after the first dose of treatment
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Groups:
- Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions): Participants with cut or subcut lesions received escalating doses of ulevostinag via IT injection on Days 1, 8, and 15 of each 21-day cycle for Cycles 1, 2, and 3 and then on Day 1 of each 21-day cycle for Cycles 4 and beyond PLUS pembrolizumab (pembro) via intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years). Note: This combination therapy treatment group includes switch-over participants from Part 1 Arm 1.
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions)
Number analyzed (Participants) | 31 | 65 | 25
Percentage of participants | 15.1 [6.6 to 21.8] | 10.4 [5.3 to 14.5] | 0 [0.0 to 6.0]

2. Primary Outcome: Parts 1 and 2: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: AEs are defined as any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study treatment, is also an AE.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC
Number analyzed (Participants) | 32 | 66 | 26 | 21 | 25
Participants | 32 | 66 | 26 | 21 | 25

3. Primary Outcome: Parts 1 and 2: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC
Number analyzed (Participants) | 32 | 66 | 26 | 21 | 25
Participants | 3 | 7 | 3 | 3 | 2

4. Secondary Outcome: Parts 1 and 2: Ulevostinag Area Under the Plasma Drug Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24)
Description: The AUC0-24 is a measure of the amount of drug in the blood over time for 0 hours to 24 hours. The AUC0-24 of ulevostinag administered via IT injection as monotherapy and the AUC0-24 of ulevostinag administered via IT injection as combination therapy with pembrolizumab IV infusion were evaluated.
Time Frame: Cycle 1 Day 1: Predose, at end of IT injection (up to 15 minutes) and 0.5, 1, 1.5, 4, 6, 12, and 24 hours postdose. Each cycle was 21 days.
Population: All participants who complied with the protocol sufficiently to ensure that the data they generated were likely to exhibit the effects of treatment, according to the underlying scientific model
Measure: Median (Full Range); unit: nM*hr
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC
Number analyzed (Participants) | 28 | 48 | 22 | 13 | 20
nM*hr | 8.62 [0.31 to 34.67] | 6.59 [0.57 to 41.43] | 5.88 [0.11 to 24.3] | 6.24 [1.78 to 12.4] | 7.98 [2.43 to 13.48]

5. Secondary Outcome: Parts 1 and 2: Ulevostinag Minimum Plasma Concentration (Cmin)
Description: Cmin is a measure of the minimum amount of drug in the plasma after the dose is given. The Cmin of ulevostinag administered via IT injection as monotherapy and the Cmin of ulevostinag administered via IT injection as combination therapy with pembrolizumab IV infusion were evaluated.
Time Frame: Cycle 1 Day 1: Predose, at end of IT injection (up to 15 minutes) and 0.5, 1, 1.5, 4, 6, 12, and 24 hours postdose; Cycle 2 Day 1: Predose, at end of IT injection (up to 15 minutes) and 0.5, 1, 1.5, 4, and 6 hours postdose. Each cycle was 21 days.
Population: as for outcome 4
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC
Number analyzed (Participants) | 28 | 48 | 22 | 13 | 20
ng/mL | 0.18 [0.06 to 3.09] | 0.12 [0.05 to 1.16] | 0.08 [0.05 to 6.83] | 0.09 [0.05 to 0.56] | 0.13 [0.05 to 0.44]

6. Secondary Outcome: Parts 1 and 2: Ulevostinag Maximum Plasma Concentration (Cmax)
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. The Cmax of ulevostinag administered via IT injection as monotherapy and the Cmax of ulevostinag administered via IT injection as combination therapy with pembrolizumab IV infusion were evaluated.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Median (Full Range); unit: nM
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC
Number analyzed (Participants) | 28 | 48 | 22 | 13 | 20
nM | 6.56 [0.15 to 49.9] | 5.38 [0.21 to 45.5] | 7.08 [0.43 to 48.9] | 6.75 [0.07 to 40.9] | 8.4 [0.92 to 23.8]

7. Secondary Outcome: Parts 1 and 2: Pembrolizumab Minimum Plasma Concentration (Cmin)
Description: Cmin is a measure of the minimum amount of drug in the plasma after the dose is given. The Cmin of pembrolizumab IV infusion in combination with MK-1454 administered via IT injection was evaluated.
Time Frame: Predose on Day 1 of Cycles 1, 2, and 4, and every 4 cycles thereafter up to Cycle 35 (up to 2 years). Each cycle was 21 days.
Population: as for outcome 4
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC
Number analyzed (Participants) | 32 | 18 | 15 | 19
ng/mL | 14.5 [5.03 to 68.3] | 14.25 [5.5 to 81.7] | 17.7 [7.09 to 43.2] | 13.6 [3.54 to 22.7]

8. Secondary Outcome: Parts 1 and 2: Objective Response Rate (ORR) As Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The ORR of ulevostinag at the preliminary RP2D in combination with pembrolizumab will be assessed by RECIST 1.1 modified to follow a maximum of 10 target lesions with a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 2 years
Population: All participants with a baseline scan that demonstrated measurable disease by investigator assessment, and who received a dose of study medicine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC
Number analyzed (Participants) | 30 | 62 | 26 | 21 | 25
Percentage of participants | 0.0 [0.0 to 11.6] | 16.1 [8.0 to 27.7] | 3.8 [0.1 to 19.6] | 4.8 [0.1 to 23.8] | 4.0 [0.1 to 20.4]

ADVERSE EVENTS:
Time Frame: Up to approximately 2 years
Description: All-Cause Mortality population includes all allocated participants. Serious and Other Adverse Events population includes all participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment are excluded as AEs.
Arm/Group | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC
All-Cause Mortality (participants affected / at risk) | 21/32 | 45/66 | 19/26 | 19/21 | 15/25
Serious Adverse Events (participants affected / at risk) | 14/32 | 33/66 | 10/26 | 11/21 | 7/25
Other Adverse Events (participants affected / at risk) | 32/32 | 65/66 | 26/26 | 21/21 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) (N=32) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) (N=66) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) (N=26) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory (N=21) | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Injection site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Product dispensing error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Arm 1: Ulevostinag (Cut/Subcut Lesions) (N=32) | Part 1 Arm 2: Ulevostinag+Pembro (Cut/Subcut Lesions) (N=66) | Part 1 Arm 3: Ulevostinag+Pembro (Visceral Lesions) (N=26) | Part 2 Cohort A: HNSCC Anti-PD-1/PD-L1 Refractory (N=21) | Part 2 Cohort B: Anti-PD-1/PD-L1 TrT-Naïve or Refractory TNBC (N=25)
Anaemia (Blood and lymphatic system disorders) | 14 (17) | 27 (42) | 6 (11) | 11 (14) | 7 (9)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (9) | 7 (8) | 5 (5) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 15 (16) | 2 (2) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (11) | 14 (26) | 2 (2) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 16 (22) | 16 (21) | 6 (10) | 8 (8) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (13) | 9 (17) | 8 (9) | 3 (3) | 1 (1)
Asthenia (General disorders) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 4 (4)
Chest pain (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 17 (55) | 24 (59) | 12 (28) | 5 (11) | 9 (19)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 17 (19) | 28 (34) | 12 (25) | 5 (8) | 3 (3)
Influenza like illness (General disorders) | 7 (11) | 15 (45) | 0 (0) | 5 (14) | 0 (0)
Injection site erythema (General disorders) | 5 (6) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 1 (1)
Injection site necrosis (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 19 (34) | 21 (46) | 6 (9) | 4 (5) | 4 (7)
Injection site reaction (General disorders) | 3 (4) | 9 (12) | 1 (1) | 1 (1) | 3 (10)
Injection site swelling (General disorders) | 3 (4) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 7 (7) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 24 (58) | 38 (85) | 20 (51) | 11 (20) | 20 (53)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 4 (9) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 7 (9) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (6) | 3 (7) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 8 (12) | 1 (1) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 11 (14) | 6 (6) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 11 (11) | 5 (5) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 1 (5)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 10 (11) | 3 (3) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 13 (14) | 9 (15) | 5 (5) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (10) | 0 (0) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (7) | 0 (0) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 8 (8) | 2 (6) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 11 (30) | 2 (3) | 2 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 5 (8) | 0 (0) | 2 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 11 (17) | 3 (3) | 2 (3) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (5) | 3 (3) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (18) | 6 (9) | 6 (9) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (16) | 0 (0) | 5 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 11 (20) | 1 (1) | 2 (2) | 1 (3)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 2 (2) | 3 (3) | 3 (3) | 2 (4)
Dizziness (Nervous system disorders) | 3 (3) | 7 (8) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (18) | 15 (28) | 4 (7) | 0 (0) | 2 (5)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 13 (15) | 2 (2) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8) | 3 (3) | 2 (2) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 8 (10) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 8 (20) | 7 (14) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 18 (23) | 5 (5) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 9 (10) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (10) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (6) | 0 (0) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 5 (5) | 9 (9) | 4 (4) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03010176/Prot_SAP_000.pdf